CLINICAL TRIAL: NCT03873376
Title: A Pragmatic Randomized Controlled Trial of Self-sampling Among Long-term Non-attenders to Cervical Cancer Screening
Brief Title: Self-sampling Among Long-term Non-attenders to Cervical Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); University of Oslo (Other); University of Bergen (Other); Albert Einstein College of Medicine (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Bo Terning Hansen, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18/14056; 182687 (Other: Cancer Society of Norway (Funder))
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Cervical Cancer
Keywords: mass screening; non-attendance; self-sampling; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opt-in (Experimental): Receive offer to order self-sampling kit
  Interventions: Behavioral: Opt-in; Receive offer to order self-sampling kit
- Opt-out (Experimental): Receive self-sampling kit unsolicited
  Interventions: Behavioral: Opt-out; Receive self-sampling kit unsolicited
- Control (Experimental): Receive open reminder to be screened by physician
  Interventions: Behavioral: Control; Receive open reminder to be screened by physician

INTERVENTIONS:
Behavioral: Opt-in; Receive offer to order self-sampling kit — Women in the opt-in arm receive an offer to order a HPV self-sampling kit, in addition to information about the study. Women who order, receive a kit that includes a self-sampling brush (Evalyn, Rovers Medical Devices), with instructions for use and a pre-paid envelope for returning the brush for HPV testing. The women are also informed that they can attend ordinary screening, i.e. performed by a physician. Women who choose self-sampling and test positive for high-risk HPV will be 1:1 allocated to follow-up by their general practitioner or a gynecologist. Women who test negative for high-risk HPV return to the ordinary screening program
  Arms: Opt-in
Behavioral: Opt-out; Receive self-sampling kit unsolicited — Women in the opt-out arm receive the self-sampling kit directly, without having ordered it themselves. The kit has the same contents, and the follow-up is the same, as that described for the opt-in arm.
  Arms: Opt-out
Behavioral: Control; Receive open reminder to be screened by physician — Similar to the procedure of the national screening program, women in the control arm receive a reminder to be screened by their general practitioner, and continues in the ordinary screening program
  Arms: Control

SUMMARY:
The trial will evaluate whether human papillomavirus (HPV) self-sampling may increase cervical cancer screening attendance among under-screened women in Norway, how different ways of offering self-sampling and follow-up may affect attendance, and whether self-sampling may reduce inequities in attendance.

DETAILED DESCRIPTION:
A randomized control trial will be performed on the effect of vaginal HPV self-sampling on screening attendance, targeting women age 35-69 who have not attended screening for at least 10 years. The women will be randomly allocated to one of three interventions: (i) receive a reminder to be screened by a physician; (ii) receive a self-sampling kit; (iii) receive an offer to order a self-sampling kit. Comparisons of the screening attendance among the interventions will be made. To also address potential effects on inequities, the analyses will include comparisons by sociodemographic characteristics. The rates of cervical cancer/precancer among the interventions will also be compared. Further, to assess the feasibility of and the compliance to follow-up after a positive HPV test in this population, half of the HPV-positive women from each self-sampling arm will be referred to initial follow-up by their regular general practitioner (GP), while the other half will be referred to initial follow-up by a gynecologist. The project will be embedded in the national cervical cancer screening program, and will utilize the extensive nationwide registers describing performance and outcomes of screening collected by the Cancer Registry of Norway.

ELIGIBILITY:
Inclusion Criteria:

* Women living in the regions Hordaland, Vest-Agder, Rogaland or Sør-Trøndelag, who have been eligible for screening in Norway, but who have not attended screening for at least 10 years (2009-2018)

Exclusion Criteria:

* Women who have not been eligible for cervical cancer screening during the entire 10 year period (2009-2018)

Ages: 35 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5669 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Screening attendance rate (%) | 6 months
  The primary outcome measure is the attendance rate to cervical cancer screening. Attendance is defined as returning a self-sampling test, or being screened by a physician during the 6 months following receipt of the invitation letter

SECONDARY OUTCOMES:
Prevalence of high-risk HPV (%) | 6 months
  Self-samples as well as physician-taken samples will be tested for high-risk HPV with the Cobas 4800 HPV-DNA test at the national HPV reference laboratory
Prevalence of CIN2+ (proportion of cervical intraepithelial neoplasia grade 2 or worse) | 6 months
  Histologically confirmed CIN2+ diagnoses of all study participants who are eligible for follow-up will be retrieved from the cervical screening registry at the Cancer Registry of Norway
Compliance to clinical follow-up of a high-risk HPV positive screening test (%) | 6 months
  Attendance to follow-up among women with a positive screening test will be surveyed following notification of the positive test result. In addition to comparing arms, we will compare compliance of women in the self-sampling arms who are followed up by their regular GP vs. women who are followed up by a gynecologist

OTHER OUTCOMES:
Sociodemographic characteristics (%) | Up-to-date sociodemographic data retrieved from national registries in 2019
  We will compare the distribution of sociodemographic characteristics (income, education, immigration status, age etc.) by intervention and attendance status

CONTACTS AND LOCATIONS:
Overall Officials: Giske Ursin, MD, Prof, Study Director — Oslo University Hospital
Locations (1):
- Cancer Registry of Norway, Oslo, Pb 5313 Majorstuen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aasbo G, Trope A, Nygard M, Christiansen IK, Baasland I, Iversen GA, Munk AC, Christiansen MH, Presthus GK, Undem K, Bjorge T, Castle PE, Hansen BT. HPV self-sampling among long-term non-attenders to cervical cancer screening in Norway: a pragmatic randomised controlled trial. Br J Cancer. 2022 Nov;127(10):1816-1826. doi: 10.1038/s41416-022-01954-9. Epub 2022 Aug 23. PMID 35995936